CLINICAL TRIAL: NCT03790215
Title: Prospective One-arm Cohort Study of Dydrogesterone in the Treatment of Endometrial Polyps
Brief Title: Dydrogesterone in the Treatment of Endometrial Polyps
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, shuwang, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-1
Record Dates: First submitted 2018-12-21; First posted 2018-12-31 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Endometrial Polyp
MeSH Terms: interventions — Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort for treatment (Experimental): Participants enrolled are given dydrogesterone tablet of 10mg twice a day, from day 15 to day 24 of the menstrual cycle over a period of 3 months.
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Dydrogesterone — The investigators give participants oral dydrogesterone(as described in arm description).After 3 cycles of treatment, the investigators evaluate the treatment effects.
  Other Names: Duphaston

SUMMARY:
This study is intended to observe the therapeutic effect of dydrogesterone on endometrial polyps and provide a reference for clinical treatment.

DETAILED DESCRIPTION:
Endometrial polyps are a common female endometrial lesion.The long-term unrestrained exposure of estrogen to local tissue is one of the causes of polyp formation.Studies suggested that the progesterone can accelerate the regression rate of endometrial polyps due to its antiestrogenic effects.Based on this, investigators intended to observe the therapeutic effect of dydrogesterone on endometrial polyps and provide a reference for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. women of childbearing age from 20 to 50 years old
2. with or without menstrual changes:

   1. menostaxis (longer than 7 days)
   2. shortened menstrual cycles(less than 23 days)
   3. menorrhagia(more than twice as much as usual)
   4. abnormal vaginal bleeding(non-menstrual vaginal bleeding)
3. with following signs of vaginal ultrasound in the follicular phase (day 1 to day 10 of a menstrual cycle):

   1. typical signs with a suspect of EP: (median/high) echo with a regular contour within the uterine lumen;
   2. atypical signs with a suspect of EP: punctate cystic areas within the endometrium and the endometrial thickness >1cm;

Exclusion Criteria:

1. no menses within half a year;
2. surgery or drug treatment of endometrial lesions in the past half year;
3. with current intrauterine device;
4. combined with other acute gynecological inflammation;
5. with clinically suspected malignant tumors;
6. long-term use of oral contraceptives;
7. with abnormal liver and kidney function;
8. with benign or malignant breast tumors;
9. with any systemic malignant tumor or a history of tumors;
10. participants who are pregnant.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Regression rate of endometrial polyps | three months after the starting of treatment
  No evidence of polyps or the maximum dimensions of polyps are reduced by 1/3 or more under pelvic ultrasound
Relapse rate of endometrial polyps | six months after the starting of treatment
  Evidence of polyps or the maximum dimensions of polyps are larger during the follow-up of the regression group after treatment

SECONDARY OUTCOMES:
Side effects | three months after the starting of treatment
  Any side effects during the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China